CLINICAL TRIAL: NCT03355378
Title: Short Versus Standard Post-operative Stay After Elective Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POSCS
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): gum chewing during spinal anesthesia and early ambulation
  Interventions: Procedure: gum chewing
- Control group (No Intervention): no gum chewing

INTERVENTIONS:
Procedure: gum chewing — chewing gum orally for 30 minutes
  Arms: study group

SUMMARY:
After major open abdominal surgery, transient paralytic ileus usually follows. It has been suggested that stimulation of pain fibers, excessive sympathetic tone, and the release of inhibitory neurotransmitters from bowel wall associated with bowel manipulation and peritoneal irritation are responsible mechanisms. There have been concerns that early postoperative oral feeding would lead to vomiting with subsequent aspiration pneumonia, anastomotic leakage, and wound dehiscence.

ELIGIBILITY:
Inclusion Criteria:

1. Women is sure of her last menstrual period or documented early pregnancy ultrasound.
2. Women aged 20-35 years.
3. Women with Body mass index18-22 kg/m2.
4. Estimated gestational age is ranging between 37-40 weeks gestation.
5. Accepting to participate in the study.

Exclusion Criteria:

1. Smoker ≥ 11 cigarettes/day.
2. Caesarean hysterectomy .
3. Surgical management of severe postpartum haemorrhage .
4. History of bowel obstruction , inflammatory bowel disease .
5. Previous abdominal or pelvic radiation

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
duration of hospital stay | 48 hours
  time of postoperative recovery of gastrointestinal tract

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt